CLINICAL TRIAL: NCT04999059
Title: A Long-Term Follow-Up Study of Subjects With Fabry Disease Who Previously Received Ex-Vivo, Lentiviral Vector-Mediated Gene-Modified Autologous Cell Therapy AVR-RD-01 in Study AVRO-RD-01-201
Brief Title: Long-Term Follow-up Study of Subjects With Fabry Disease Who Received Lentiviral Gene Therapy in Study AVRO-RD-01-201
Status: Terminated | Type: Observational
Why Stopped: This study was voluntarily terminated due to a business decision not to proceed, and not due to any safety or efficacy issue.
Sponsor: AVROBIO (Industry)
Responsible Party: Sponsor
Other Study IDs: AVRO-RD-01-LTF01
Record Dates: First submitted 2021-08-04; First posted 2021-08-10 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2022-10

CONDITIONS: Fabry Disease
Keywords: Fabry Disease; Cell therapy; Gene therapy; Long-term follow-up; Lysosomal storage disorder; Lenti-viral
MeSH Terms: conditions — Fabry Disease; Lysosomal Storage Diseases | interventions — Safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample collections including serum chemistry (and electrolytes), hematology, and anti-AGA antibodies, and urinalysis. Bone marrow aspirate for efficacy, and reproductive testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Fabry Disease: This is a long-term follow-up study of participants who previously received AVR-RD-01 (single dose administration) in the AVRO-RD-01-201 treatment study. No investigational product will be administered in this study.
  Interventions: Other: Safety and Efficacy Assessments

INTERVENTIONS:
Other: Safety and Efficacy Assessments — Safety evaluations, disease-specific assessments, and other assessments to monitor for long-term complications of gene therapy intervention.
  Other Names: Gene Therapy Intervention

SUMMARY:
This is a multinational, long-term follow-up study to assess the long-term safety and durability of AVR-RD-01 treatment in participants who received a single dose administration of lentiviral gene therapy in Study AVRO-RD-01-201 (treatment study). No investigational product will be administered in this study. Participants will continue periodic safety and efficacy assessments in this long-term follow-up study up to 15 years from AVR-RD-01 gene therapy infusion.

DETAILED DESCRIPTION:
Participants enrolled in the AVRO-RD-01-201 study will be offered participation in the AVRO-RD-01-LTF01 study. The Baseline visit for the AVRO-RD-01-LTF01 study will coincide with the participant's last visit in the AVRO-RD-01-201 study. Participants confirmed eligible for the AVRO-RD-01-LTF01 study will be asked to return for study visits at approximately 6-month intervals for the first 4 years and annually thereafter for 10 years (for a total of 15 years from AVR-RD-01 infusion) during which time continued safety, engraftment, and efficacy of treatment will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have been enrolled and received AVR-RD-01 in the AVRO-RD-01-201 study.

Exclusion Criteria:

1. Subject has any medical, psychological, or other condition that, in the opinion of the Investigator:

   * Might interfere with the subject's participation in the study (including consenting to procedures); and/or
   * Poses any additional risk to the subject; and/or
   * Might confound the results of any study-required assessments.
2. Subject is currently enrolled in an AVROBIO-sponsored AVR-RD-01 treatment study.

Ages: 16 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects who received AVR-RD-01 in the preceding treatment study, meet all eligibility criteria, and agree to comply with the study visit schedule and procedures.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
Incidence of clinically significant AEs and SAEs | Baseline to Year 15 post gene therapy infusion
Number of participants with clinically relevant abnormalities, as assessed by clinical laboratory tests | Baseline to Year 15 post gene therapy infusion
Number of participants with clinically relevant abnormalities, as assessed by vital signs | Baseline to Year 15 post gene therapy infusion
Presence of anti-Alpha-galactosidase A (AGA) antibodies | Baseline to Year 15 post gene therapy infusion
Presence of replication competent lentivirus (RCL) | Baseline to Year 15 post gene therapy infusion
Evaluate for the presence of aberrant clonal expansion as assessed by integration site analysis (ISA) | Baseline to Year 15 post gene therapy infusion

SECONDARY OUTCOMES:
Change from baseline in AGA enzyme activity level and peripheral blood leukocytes (PBLs) | Baseline to Year 15 post gene therapy infusion
Average Vector Copy Number (VCN) in peripheral blood leukocytes as assessed by quantitative polymerase chain reaction (qPCR) and/or droplet digital polymerase chain reaction (ddPCR) | Baseline to Year 15 post gene therapy infusion
Change from baseline in Globotriaosylceramide (Gb3) biomarkers for Fabry disease in plasma and urine | Baseline to Year 15 post gene therapy infusion
Average Vector Copy Number (VCN) in bone marrow / progenitor cells as assessed by quantitative polymerase chain reaction (qPCR) and/or droplet digital polymerase chain reaction (ddPCR) | Baseline to Year 15 post gene therapy infusion
Change from baseline in eGFR | Baseline to Year 15 post gene therapy infusion
Change from baseline in left ventricular mass index (LVMI) as assessed by cardiac magnetic resonance imaging (MRI) | Baseline to Year 15 post gene therapy infusion
Change from baseline in abdominal pain and stool consistency as assessed by the Diary for Irritable Bowel Syndrome Symptoms-Diarrhea (DIBSS-D) | Baseline to Year 15 post gene therapy infusion
Change from baseline in Brief Pain Inventory-Short Form (BPI-SF) questionnaire scores | Baseline to Year 15 post gene therapy infusion
Change from baseline in physical and mental functioning as assessed by the Short Form 36 (SF-36) Physical Component Summary (PCS) and Mental Component Summary (MCS) scores | Baseline to Year 15 post gene therapy infusion

CONTACTS AND LOCATIONS:
Overall Officials: Inderpal Panesar, MRPharmS, Study Director — AVROBIO, Inc
Locations (3):
- Australia (2):
  - Royal Melbourne Hospital, Melbourne, Parkville VIC
  - Royal Perth Hospital, Perth
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil